CLINICAL TRIAL: NCT07363551
Title: Omega-3 Fatty Acids, Inflammation, Gut Microbiota in Youth With Depression (OMIMYDep)- A Double-blind Randomized Controlled Trial
Brief Title: Omega-3 Fatty Acids, Inflammation, Gut Microbiota in Youth With Depression
Acronym: OMIMYDep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Pei-Chen Chang, Consultant Psychiatrist, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC3-129
Record Dates: First submitted 2024-04-25; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ADHD
Keywords: omega-3, ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: To investigate the effects of omega-3 in youth with depression
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 (Active Comparator): EPA
  Interventions: Combination Product: Omega-3 fatty acids
- placebo (Placebo Comparator): soy bean oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Combination Product: Omega-3 fatty acids — omega-3 fatty acids (EPA)
  Arms: omega-3
Dietary Supplement: Placebo — soy bean oil
  Arms: placebo

SUMMARY:
This is a 12 week double blind RCT aimed to investigate the role of omega-3 fatty acids in patients with major depressive disorder

DETAILED DESCRIPTION:
This is a 12 week double blind RCT aimed to investigate the role of omega-3 fatty acids in patients with major depressive disorder. Outcome measures including clinical symptoms, inflammation biomarkers and gut microbiota profiles.

ELIGIBILITY:
Inclusion Criteria:

* Youth with a DSM-5 diagnosis of MDE

Exclusion Criteria:

* Has a recent change in antidepressants or psychotherapy treatment within 4 weeks.
* Allergic to omega-3 fatty acids

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
clinical symptoms | week 0,1,2,4,8,12
  Hamilton Depression Rating Scale (HAMD)-21 item is a clinician-rated scale designed to assess the severity of depressive symptoms over the past week. It is commonly used in clinical trials and psychiatric practice Total Score Interpretation (Commonly Used) Total Score and Severity Level
  * 0-7: No depression / Normal
  * 8-13: Mild depression
  * 14-18: Moderate depression
  * 19-22: Severe depression -≥23: Very severe depression

SECONDARY OUTCOMES:
gut microbiota | week 0,12
  gut microbiota
inflammatory cytokines (IL-6, hsCRP) | week 0,12
  blood inflammatory cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taichung, Taiwan